CLINICAL TRIAL: NCT05224622
Title: Detection of the 2019 Novel Coronavirus (SARS-CoV-2) Using Breath Analysis - Validation Study.
Brief Title: Detection of COVID-19 Using Breath Analysis - Validation Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scentech Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COV-2-PMC-2021
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drive In (Experimental): Drive In attendees will undergo one breath sampling.
  Interventions: Diagnostic Test: VOX
- Healthy (Experimental): Healthy attendees will undergo two successive breath sampling.
  Interventions: Diagnostic Test: VOX
- Corona Department (Experimental): Healthy attendees will undergo five successive breath sampling.
  Interventions: Diagnostic Test: VOX

INTERVENTIONS:
Diagnostic Test: VOX — Breath exhalation into the mouthpiece of the VOX breath diagnostic device.

SUMMARY:
Detection of the 2019 novel Coronavirus (SARS-CoV-2) using breath analysis - Validation study.

DETAILED DESCRIPTION:
A diagnostic prospective single-site study, with no anticipated risks or constraints.

Primary objective- To validate the value of a set of breath VOC biomarkers that enable the investigator to distinguish between COVID-19 carriers and COVID-19 non-carriers in comparison to the gold-standard testing methodology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years at the time of consent
* Capable of understanding written and/or spoken language
* Able to provide informed consent
* Was not treated with Anti-viral drugs

Exclusion Criteria:

* Age under 18 years old
* Under guardianship or deprived of liberty
* Pregnant or lactating woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Presence of Volatile Organic Compounds indicating carriers of COVID-19. | Through the study completion, up to 3 months.
  Obtain early verification accuracy of measures for a set of VOCs biomarkers indicating carriers of Corona virus.

SECONDARY OUTCOMES:
Association of exhaled biomarkers with participants' characteristics (age, gender, symptoms-severity, etc.) | Through the study completion, up to 3 months.
  Correlation level between exhaled biomarkers and participants' demographic characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Peretz, PhD, Principal Investigator — Poriya Medical Center
Locations (1):
- Poriya Medical Center, Poria – Neve Oved, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD